CLINICAL TRIAL: NCT01411046
Title: Observational Cohort Study on Difference in Glucocorticoid-induced Adrenal Insufficiency in Patients With Rheumatoid Arthritis Related to Different Sensitivity Polymorphisms in the Glucocorticoid Receptor Gene
Brief Title: Difference in GC-induced Adrenal Insufficiency in RA Related to Polymorphisms in the Glucocorticoid Receptor Gene
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulla Feldt-Rasmussen, Professor, Rigshospitalet, Denmark
Other Study IDs: GCR-RA-CSI
Record Dates: First submitted 2011-07-28; First posted 2011-08-05 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Glucocorticoid; polymorphism; Glucocorticoid receptor gene; rheumatoid arthritis; adrenal insufficiency; prednisolone treatment
MeSH Terms: conditions — Arthritis, Rheumatoid; Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples and DNA from gene analyses
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- RA treated with prednisolone: Patients with RA treated with prednisolone, minimum 5 mg/day for minimum 6 months. Patients are grouped according to haplotype of 4 SNPs of the glucocorticoid recepror gene. Patients with or without these polymorphisms were invited to a Synacthen® test, but patients with a mixed hetero- and homozygote genotype were not. Adrenal function is evaluated with a Synacthen test.
  Interventions: Diagnostic Test: Synacthen test

INTERVENTIONS:
Diagnostic Test: Synacthen test — 250 microg Synacthen test, performed fasting, in the morning, starting between 08·00 and 10·30 h, after an overnight fast and a prednisolone pause of approximately 48 hours (depending on normal dose administration time).

SUMMARY:
Development of glucocorticoid (GC)-induced adrenal insufficiency is a serious adverse effect of GC treatment. It is today not possible to predict this adverse effect. The project aims at investigating a possible individual aspect, which may render subjects more or less sensitive to glucocorticoids, and thereby influence development of GC induced adrenal insufficiency. The hypothesis is that subjects with one or another of the polymorphisms in the GC receptor gene will either have increased or diminished GC sensitivity. This may be responsible for differences in development of GC induced adrenal insufficiency.

DETAILED DESCRIPTION:
Blood is sampled from patients with rheumatoid arthritis (RA), fulfilling the inclusion criteria and patients are genotyped for the SNPs N363S, BclI, ER22/23EK and 9β and grouped according to haplotypes. SNPs will be determined by polymerase chain reaction (PCR). Patients will be included for a Synacthen test, to evaluate their adrenal function. Information from the results of the study will be able to assist clinicians to identify patients at risk and thus individualize GC therapy in a tailored fashion. Results of the study will be important for all patient groups worldwide on GC therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years)
* Caucasian classified with rheumatoid arthritis.
* 1987 ACR-classification criteria.
* Prednisolone min 5mg/day for at least 6 months.
* Presence of either BclI (high GC sensitivity) or 9β (low GC sensitivity)polymorphisms, or wildtype for for all 4 SNPs studied. Patients with or without these polymorphisms were invited to a Synacthen® test, but patients with a mixed hetero- and homozygote genotype were not

Exclusion Criteria:

* Other major organ disease
* Females pregnant
* Females not willing to pause estrogen-containing medications 6 weeks prior to Synacthen® test
* unable to give a written informed content

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with rheumatoid arthritis in prednioslone treatment, screened for four specific polymorphisms of the glucocorticoid receptor gene.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2011-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
adrenal insufficiency | upon first visit within average 1 month
  test for adrenal function by stimulation test (Synacthen test)

SECONDARY OUTCOMES:
quality of life | upon inclusion (baseline)
  test by questionnaires
Bone Density status | results from latest DXA scan performed in routine settings, bonemarkers upon inclusion (baseline)
  DXA and bone markers
body composition | upon inclusion (baselline)
  BMI, waist-, hip- circumferencia
metabolic syndrome | upon inclusion (baseline)
  blood lipids, abdominal obesity, blood pressure, fasting plasma glucose

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided